CLINICAL TRIAL: NCT02153619
Title: Development of Psychotherapeutic Interventions for Parents Who Lost a Child
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: University of Memphis (Other); University of Hawaii (Other); Adelphi University (Other); Weill Medical College of Cornell University (Other); University of Southern California (Other); The New School for Social Research (Other); Monash University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-102
Record Dates: First submitted 2014-05-22; First posted 2014-06-03 (Estimated); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Parents Who Have Lost a Child
Keywords: Grief; bereavement; questionnaires; therapy sessions; 14-102

ARMS (2):
- Meaning-Centered Grief Therapy (MCGT) (Experimental): Part 1: Open Trials. Participants (n = 5 for Step 1 & n = 5 for Step 2) will receive 16 1-hour (approx) weekly sessions MCGT, & all therapy sessions will be audio recorded. Will make every effort to complete 16 sessions in 16 weeks, due to normal life activities, this is considered an approximation (i.e. there may be weeks where sessions don't take place &/or weeks where more than 1 session takes place in a week). If participant provides us with permission, we will also video record the sessions. Assessments will be administered at 4 time points: pre-intervention (T1), mid-intervention (T2), post-intervention (T3), & at 3-months post-intervention (T4). They will provide their feedback about MCGT & the measures. PI will review the open trial sessions to help refine the MCGT manual & treatment integrity forms. Sessions for Step 1 participants in Part 1 will be held at the MSK Counseling Center. Sessions for Step 2 participants in Part 1 will be conducted via videoconferencing.
  Interventions: Behavioral: Meaning-Centered Grief Therapy (MCGT); Behavioral: questionnaires assessments
- MCGT or Supportive Psychotherapy (Experimental): Part 2: Pilot RCT. Will randomize 66 parents to 16 weekly 60-90 minute (approx) sessions of MCGT or SP delivered via videoconferencing. Again, sessions will be audio recorded. If the participant provides us with permission, we also audio/video record the sessions. We will examine aspects of study implementation & therapy process, including a) recruitment progress, b) implementation of the intervention, c) administration of the assessments, & d) retention. We will also examine acceptability, defined as measures of satisfaction at T3. Psychosocial outcomes will be assessed with self-report measures at 4 time points: pre-intervention (T1), mid-intervention (T2), post-intervention (T3), & at 3-months post-intervention (T4). Post-intervention qualitative exit interviews will assess acceptability of the intervention. Post-intervention qualitative exit interviews will assess acceptability of the MCGT intervention .
  Interventions: Behavioral: Meaning-Centered Grief Therapy (MCGT); Behavioral: Supportive Psychotherapy (SP); Behavioral: questionnaires assessments

INTERVENTIONS:
Behavioral: Meaning-Centered Grief Therapy (MCGT) — MCGT is a manualized, one-on-one intervention that uses psychoeducation, experiential exercises, and homework focusing on themes related to meaning, identity, purpose, and legacy. Post-intervention qualitative exit interviews will assess acceptability of the MCGT intervention (see Appendix I). Participants randomized to MCGT will provide their feedback about MCGT and the measures (n = 33).
Behavioral: Supportive Psychotherapy (SP) — "SP is the comparison condition in this study and is a standardized, manualized intervention developed by the MSK Psychiatry Service and utilized in our completed and ongoing RCTs of Meaning-Centered Psychotherapy."
  Arms: MCGT or Supportive Psychotherapy
Behavioral: questionnaires assessments

SUMMARY:
Many parents who have lost a child use counseling or other resources to help with the emotional burden of their loss. The aim of this study is to begin to test a new counseling program for parents who have lost a child.

DETAILED DESCRIPTION:
There are two parts to this study. Adapting and refining the MCGT intervention manual will be accomplished primarily in Part 1, building upon a preparatory project to obtain feedback on the MCGT intervention manual and materials.

Step 1 of Part 1 will involve a brief open trial of MCGT delivered in person at an MSK location with individual parents (n=5) to further refine the treatment through active participant feedback and identify ways to improve therapeutic alliance to maximize the impact of delivery via videoconferencing. Parents may also invite a support provider to join them for Session 9 (support provider n = 5). Support providers will not be evaluated as research participants.

Step 2 of Part 1 will be another brief open trial (n=5) delivering MCGT via video conferencing to iron out any logistical challenges prior to the pilot randomized controlled trial (RCT). The investigators hope to use videoconferencing in order to ultimately improve parents' access to supportive services. Participants will be able to complete sessions wherever they have both privacy and access to a computer and the internet. Parents may also invite a support provider to join them for Session 9 (support provider n = 5). Support providers will not be evaluated as research participants.

All Part 1 participants will be assessed pre-intervention (T1), mid-intervention (T2), post-intervention (T3), and at 3-months post-intervention (T4). A qualitative exit interview will also be conducted post-intervention. This interview will be audio recorded. Video recording of the exit interview will be optional. Throughout both steps, parent testimonials that address barriers to accessing mental health services will be obtained to assist in Part 2 outreach and recruitment.

Part 1 will be conducted with parents experiencing elevated PGD symptoms as measured by the PG-13, a 13-item self-report scale evaluating PGD symptom severity, duration, and impairment. For this study, PG-13 scores ≥ 34 will be considered indicative of elevated PGD symptoms.

Part 2 will be used to obtain information about the feasibility, tolerability, acceptability, and effect size estimates of MCGT (delivered via video conferencing) to assist in planning a larger, efficacy RCT. These goals will be accomplished by undertaking a parallel-arm RCT comparing the refined MCGT to a standardized supportive psychotherapy (SP), both one-on-one interventions delivered via videoconferencing, which numerous studies show is as efficacious as in-person delivery.15-17 Parents (n=56) with PG-13 scores ≥ 34 will be randomized to receive MCGT or SP to compare their relative feasibility, acceptability, tolerability, and preliminary effects. As in Part 1, participants will be assessed pre-intervention (T1), mid-intervention (T2), post-intervention (T3), and at 3-months post-intervention (T4). All psychotherapy sessions for Part 1 will need to be completed before Part 2 begins. The investigators expect that they will be able to begin Part 2 of the protocol (during which recruits 56 parents) approximately 3 months after the final parent is enrolled in Part 1, Step 2. Approximately 56 parents (individuals) will complete the intervention in Part 2.Parents randomized to MCGT may also invite a support provider to join them for Session 9 (support provider n = 28). Support providers will not be evaluated as research participants. 1-2 training cases per MCGT interventionist (rather than randomized) will also be enrolled on this study for training purposes. There may be weeks where sessions do not take place and/or weeks where more than one session takes place in a week.

Past participants on the study may also be contacted to join a Parent Advisory Board (PAB) Potential members of PAB may also be identified from the community. Members of the PAB will be invited to provide their perspectives, ideas, and feedback on the intervention and ongoing and future research.

ELIGIBILITY:
Inclusion Criteria:

* Loss of a child at least 6 months
* Biological or adoptive parent or stepparent as reported in the child's medical record or by parent report
* Parent must be age 18 or over as reported by parent
* In the judgment of investigators/consenting professionals, able to comprehend English to complete study assessments
* Score of 34 or greater ( ≥ 34) on the PG-13 at screening (N/A for training case participants)
* Residing in New York, New Jersey, Connecticut, or Pennsylvania for P1S1; Residing in New York for P1S2; residing in New York or New Jersey or able to complete sessions while complying with current telehealth regulations.

Support Provider Inclusion Criteria:

* Must be age 18 or over as indicated by self-report
* Has been identified by the bereaved parent participant as a support or someone important to bereaved parent
* Must reside in New York or New Jersey or able to complete sessions while complying with current telehealth regulations.

Exclusion Criteria:

* Significant psychiatric disturbance sufficient, in the investigator's judgment, to preclude completion of the assessment measures, interview or informed consent
* Inability to access a computer with Internet or inability to use a computer with Internet provided by the study as indicated by self-report
* Another parent or primary caregiver of the child has been enrolled in the study (N/A for training case participants)
* For the Part 2 RCT, participated in Part 1, Step 1 or 2.

Support Provider Exclusion Criteria:

* Significant psychiatric disturbance sufficient, in the investigator's judgment, to preclude completion of the assessment measures, interview or informed consent
* Inability to access a computer with Internet or inability to use a computer with Internet provided by the study as indicated by self-report

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
feasibility defined and measured as the proportion of participants who complete at least 8 out of 16 sessions of therapy as well as completion of the T3 PG-13 assessment | 4 years
psychological outcome data in prolonged grief symptoms, assessed with the PG-13 summary score. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Talia Zaider, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

DOCUMENTS (1):
  • Informed Consent Form (2021-04-07): https://cdn.clinicaltrials.gov/large-docs/19/NCT02153619/ICF_000.pdf